CLINICAL TRIAL: NCT05213598
Title: Natural History of Fontan Associated Liver Disease and the Evaluation of Biomarkers for Disease Severity Assessment
Brief Title: Fontan Associated Liver Disease and the Evaluation of Biomarkers for Disease Severity Assessment
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000494; 000494-DK
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10-16

CONDITIONS: Congenital Heart Disease
Keywords: Cardiac Hepatopathy; Natural History
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with FALD: male and female subjects =18 years of age who historically underwent Fontan procedure due to a severe CHD and thus are at risk for FALD by virtue of their altered physiology

SUMMARY:
Background:

In Fontan Associated Liver Disease (FALD), congestion of blood in the liver causes cirrhosis. This condition can cause death. Researchers want to understand what triggers this process and find new treatments for it.

Objective:

To understand how long-term congestion of blood in the liver causes liver scarring that eventually leads to cirrhosis.

Eligibility:

People aged 18 and older who are at risk of developing FALD from the Fontan procedure.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Liver ultrasound. This uses sound waves to take pictures of the body.

Participants will have an outpatient visit within 12 weeks after screening. Within 24 weeks later, they will have a 3-day hospital stay. About 2 weeks later, they will have a follow-up visit.

Visits will include repeats of the screening tests and:

Heart tests

Stool collection

Questionnaires

MRI of the liver. Participants will lie on a bed that slides in and out of the scanner. They will receive a contrast agent injected into a vein. While in the scanner, they will also have an MRCP to view the bile ducts and the pancreatic duct.

Fibroscan exam. This is an ultrasound that uses a special probe to look at the toughness of the liver.

Upper endoscopy. This uses a thin scope to look inside the upper digestive tract.

Liver biopsy. This will be taken through large vein in the neck or through the chest. Just before the biopsy, participants will have pressure measurements inside their liver. For this, a catheter will be inserted into a neck vein and guided into the liver.

DETAILED DESCRIPTION:
Study Description:

Up to 100 subjects who completed the Fontan procedure for severe Congenital Heart Disease (CHD) and are at risk for congestive hepatopathy or Fontan Associated Liver Disease (FALD) will be offered inclusion in the study. During the study we will pursue novel biomarkers for disease severity.

Objectives:

Primary Objective:

The goal of this study is to globally investigate a large cohort of FALD subjects to generate an understanding of how congestive hepatopathy drives the pathogenesis of cirrhosis in FALD. We will use our findings to generate novel biomarkers that will enable improved follow-up of subjects and enhance transplant decision making.

Secondary Objectives:

1. Measurement of TGF-beta serum levels in Fontan subjects and comparing them to liver tissue biopsies in hope of pursuing a novel biomarker for the development of advanced FALD.
2. Evaluation of FALD subjects coagulation profile including von Willebrand factor assessment and correlating it to disease severity by liver biopsy.
3. Comparison of PAR-1 and PAR-2 receptor staining from liver tissue biopsies of Fontan subjects and corelate their presence to the severity of the subjects FALD.
4. Identification of genetic modifiers of FALD
5. Evaluation of hepatic transcriptome in various stages of FALD.
6. Characterization of microbiome signatures in FALD

Endpoints:

Primary Endpoints:

1. Identification of novel biomarkers correlating with disease progression markers in Fontan Associated Liver Disease.
2. Develop an understanding of the biological mechanisms and the genetic modifiers of the progression of Fontan Associated Liver Disease.

Secondary Endpoints:

1. TGF-beta superfamily measurement in serum and establishment of a cut-off level correlating with FALD severity.
2. Complete coagulation profile measurement and vWF-Ag quantification with establishment of cut- offs correlating with FALD severity.
3. PAR-1 and PAR-2 immuno-staining in Fontan subjects liver tissue biopsies.
4. Establishment of positive or negative correlation between candidate susceptible genes and disease phenotype.
5. Identification of novel markers of fibrosis or the development of hepatic neoplasia from transcriptome analysis.
6. Characterization of microbiome signatures (taxonomic and functional), as well as identification of specific species.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male and female subjects >= 18 years of age.
2. Past surgical history of Fontan procedure.
3. Prior enrollment in the Liver Diseases Branch protocol 91DK0214
4. Underwent cardiac catheterization or transjugular liver biopsy within ten years prior to the date of screening
5. Approved to proceed by the NIH Cardiology Consult
6. Approved to proceed by the NIH Cardiac Pre-anesthesia Consult

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Evidence of other forms of liver disease that typically result in cirrhosis.
2. Evidence of active Chronic Hepatitis B infection as defined by the presence of hepatitis B surface antigen (HBsAg) in serum and elevated HBV DNA (>10,000 IU/mL).
3. Hepatitis C as defined by the presence of hepatitis C RNA in serum.
4. Evidence of other liver disease such as primary sclerosing cholangitis, primary biliary cirrhosis, Wilson s disease, autoimmune hepatitis as defined by either liver histology or laboratory abnormalities.
5. Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy or homozygosity for C282Y. Patients with iron saturation indices of >45% and serum ferritin levels of >300 ng/ml for men and >250 ng/ml for women will undergo genetic testing for hemochromatosis.
6. Bile duct obstruction as suggested by imaging studies done within the previous six months.
7. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year (assessed during patient interviews or by patient self-report).
8. Evidence of hepatocellular carcinoma; either alpha-fetoprotein (AFP) levels greater than 50 ng/ml (normal <6.6 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.
9. Evidence of Cholangiocarcinoma.
10. A documented or otherwise stated severe allergic reaction to contrast.
11. Any other severe condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.
12. Radiation exposure exceeds 5 rems during the past year.
13. Inability to comply or give written informed consent as there is no direct benefit from participation in this study.
14. Female subjects who are currently pregnant will be excluded due to radiation exposure necessary for study completion. In addition, altered hemodynamics may confound the study s results. Following pregnancy, patients may be reconsidered for the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female subjects >=18 years of age who historically underwent Fontan procedure due to a severe CHD and thus are at risk for FALD by virtue of their altered physiology
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2051-06-30 (Estimated); Study Completion 2051-06-30 (Estimated)

PRIMARY OUTCOMES:
To generate understanding of how congestive hepatopathy drives the pathogenesis of cirrhosis in FALD | End of Study
  Identification of novel biomarkers correlating with disease progression markers in Fontan Associated Liver Disease Develop an understanding of the biological mechanisms and the genetic modifiers of the progression of Fontan Associated Liver Disease

SECONDARY OUTCOMES:
Comparison of PAR-1 and PAR-2 receptor staining from liver tissue biopsies of Fontan patients and corelate their presence to the severity of the patients FALD | End of Study
  PAR-1 and PAR-2 immuno-staining in Fontan subjects liver tissue biopsies
Characterization of microbiome signatures in FALD | End of Study
  Characterization of microbiome signatures (taxonomic and functional), as well as identification of specific species
Evaluation of hepatic transcriptome in various stages of FALD | End of Study
  Identification of novel markers of fibrosis or the development of hepatic neoplasia from transcriptome analysis
Identification of genetic modifiers of FALD | End of Study
  Establishment of positive or negative correlation between candidate susceptible genes and disease phenotype
Measurement of TGF-? serum levels in Fontan subjects and comparing them to liver tissue biopsies in hope of pursuing a novel biomarker for the development of advanced FALD. | End of Study
  TGF-beta superfamily measurement in serum and establishment of a cut-off level correlating with FALD severity
Evaluation of FALD patients coagulation profile including von Willebrand factor assessment and correlating it to disease severity by liver biopsy | End of Study
  Complete coagulation profile measurement and vWF-Ag quantification with establishment of cut- offs correlating with FALD severity

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this research for future research as follows: De-identified data in an NIH-funded or approved public repository@@@@@@@@@@@@Data will be shared through: An NIH-funded or approved public repository.
Supporting Information: Study Protocol
Time Frame: Date will be shared at the time of publication or shortly thereafter.
Access Criteria: PI will review requests for and approve outside collaborators under appropriate individual agreements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000494-DK.html